CLINICAL TRIAL: NCT01987921
Title: Assessment of Worldwide AKI in Pediatrics, Renal Angina and Epidemiology
Brief Title: Observational Study of Pediatric Acute Kidney Injury, Risk Factors and Outcomes
Acronym: AWARE
Status: Completed | Type: Observational
Sponsor: Children's Hospital Medical Center, Cincinnati (Other)
Responsible Party: Principal Investigator, Rajit Basu, MD MS FAAP FCCM, Co-Director, Center for Acute Care Nephrology, Children's Hospital Medical Center, Cincinnati
Other Study IDs: Pediatric AWARE Study
Record Dates: First submitted 2013-11-13; First posted 2013-11-20 (Estimated); Last update posted 2016-09-27 (Estimated); Status verified 2016-09

CONDITIONS: Acute Kidney Injury
Keywords: Acute kidney injury; Pediatrics; Critical Care
MeSH Terms: conditions — Acute Kidney Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 28 Days
Biospecimen Retention: Samples Without DNA — Urine samples will be collected from participating centers (pending local IRB approval)
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Pediatric Intensive Care Unit Patients: All patients will be included in a single cohort initially (admission to the PICU) and then cohorted into groups based on development of severe AKI (Stage 2-3 KDIGO by either Cr or UOP criteria) within the first seven days, renal angina risk strata, medical admission diagnoses, and outcomes.

SUMMARY:
Pediatric acute kidney injury (AKI) is associated with increased morbidity and mortality in critically ill patients. Currently, understanding of the epidemiology and diagnosis of AKI in children is limited by single center retrospective data and inconsistent diagnostic and stratification criteria. The hypotheses of the AWARE study is that 1) renal angina, a composite of early injury signs and risk of disease, will predict severe subsequent AKI in critically ill children and 2) the incorporation of urinary biomarkers into the renal angina scoring system will improve the prediction of the severe injury. The AWARE study is conducted to describe AKI epidemiology in a heterogeneous multinational cohort of critically ill children, characterize AKI risk factors and associated morbidity, and validate the KDIGO AKI criteria as a predictor of pediatric AKI outcomes. The multi-center, multi-national registry will create the largest ever repository of information available on AKI in children.

DETAILED DESCRIPTION:
The AWARE study is a multicenter prospective observational study designed to achieve the following three goals:

1. Establish the first international pediatric AKI registry to describe in detail the epidemiology and outcome of AKI in different pediatric and cardiac ICUs around the world.
2. Validate the precision of RAI in ruling out AKI in a large, heterogeneous study population.
3. Evaluate the predictive value of using RAI before and after the incorporation of four different urinary AKI biomarkers used in different combinations.

To achieve these primary goals, children admitted to PICUs and/or pediatric cardiac ICUs from different US and international centers will be screened for enrollment eligibility. Patients admitted to general PICU and non-surgical patients admitted to cardiac ICUs are considered the target population of AWARE. Patients admitted to neonatal ICUs and post-surgical admissions to cardiac ICUs are not included in AWARE. Both clinical variables and urinary biomarkers would be needed to accomplish the analysis.

A- Clinical variables: Clinical data of interest at study entry will include age, gender, race, ethnicity, height, weight, date of ICU admission, date of ICU discharge, date of hospital discharge, admission diagnosis(es) and primary co-morbidities. Creatinine clearance (eCrCl) will be estimated by the modified Schwartz formula29. Baseline creatinine will be collected if the patient had a listed value in the medical record in the 90 days prior to admission, with the lowest value selected if multiple measurements are present. In cases where no baseline data is available, reference eCrCl will be estimated as 120 mL/min/1.73m2. 30

Clinical data will be recorded on admission and on a daily basis for the first seven days of the PICU admission or till discharge from the PICU whatever is earlier. Another set of data will be collected to evaluate the primary and secondary outcomes of the study (see later). The outcomes data will be collected on day 28 after ICU admission when available or by most recent available data before hospital discharge for patients with no available data on day 28.

Clinical parameters of interest include:

* use of fluid resuscitation in peri-ICU period ( normal saline, PlasmalyteTM ,Ringer's Lactate, 5% Albumin, starch based fluids including dextran composites)
* daily first shift heart rate (beats per minute) from day 1 through day 7 (at the most) of ICU admission
* daily first shift respiratory rate (breaths per minute) from day 1 through day 7 (at the most) of ICU admission
* daily first shift systolic and diastolic blood pressure and mean arterial pressure (arterial line measurements will be used when available) from day 1 through day 7 (at the most) of ICU admission
* daily first shift temperature from day 1 through day 7 (at the most) of ICU admission
* use of mechanical ventilation (yes/no)
* daily first shift mean airway pressure when applicable from day 1 through day 7 (at the most) of ICU admission
* duration of mechanical ventilation
* daily first shift oxygen blood saturation ( SpO2) from day 1 through day 7 (at the most) of ICU admission
* daily first shift fraction of inspired oxygen (FiO2) (%) from day 1 through day 7 (at the most) of ICU admission
* use of nephrotoxins (yes/no) from day 0 through day 7 (at the most) of ICU admission
* types of nephrotoxic agents:

  * Nonsteroidal anti-inflammatory drugs (NSAIDS)
  * Aminoglycosides,
  * anti-viral therapy,
  * Vancomycin,
  * Piperacillin/Tazobactam,
  * Calcineurin inhibitors,
  * IV radio-contrasts ( Including Gadolinium for MRI)
* use of vasoactive support (yes/no) from day 0 through day 7 (at the most) of ICU admission
* use of diuretics on day 0 and during admission (yes/no)
* class of diuretics used (Loop diuretics, Thiazides, Potassium sparing, Carbonic anhydrase inhibitors, Vasopressin antagonist, Osmotic diuretic,)
* serum creatinine (SCr) (mg/dl) from 3 months prior to ICU admission through up 28 days after admission
* fraction of inspired oxygen (FiO2) (%) from day 1 through day 7 (at the most) of ICU admission
* total fluid in (mL) from day 0 through day 7 (at the most of ICU admission)
* total fluid out (mL) from day 0 through day 7 (at the most of ICU admission)
* total urine output (mL) from day 0 through day 7 (at the most of ICU admission)
* urine output per 12-hour shift (mL/hr) from day 0 through day 7 (at the most of ICU admission)
* use of renal replacement therapy (RRT) (yes/no)
* modality of RRT when available
* use of ventricular assisted devices or extracorporeal Membrane Oxygenation (ECMO)
* outcome data

  * mortality
  * PICU length of stay
  * hospital length of stay

Calculated daily values include:

* Change from baseline creatinine calculated as = Daily Cr/Baseline Cr
* AKI stage per Kidney Disease Improving Global Outcomes (KDIGO) guidelines

  * Stages 1,2 ,3 assessed by both creatinine and urine output (Table-1)31
  * % Fluid overload: cumulative PICU fluid overload percentage (% FO), calculated as = ((total PICU Fluid in (L) - total PICU fluid out (L)) / PICU admit weight (kg))*100
* urine output per kg per 8 hour interval
* Renal angina index (RAI) will be assessed on Days 0 and 1.
* RAI = composite of risk strata and AKI clinical injury score

  o Risk strata (AKI risk tiers):
* 1 (moderate risk): This stratum include all patients admitted to PICU and not fulfilling the criteria of high risk or very high risk strata
* 3 (high risk): This include all patients with history of solid organ or bone marrow transplantation (BMT)
* 5 (very high risk): This include all patients who receive both invasive mechanical ventilatory support AND vasoactive medication at any time in the first 12 hours of ICU admission.

  o AKI Clinical Injury scores:
* 1 (ICU status and no increase from baseline creatinine or <5% fluid overload FO)
* 2 (> 5% FO or change from baseline creatinine of 1-1.49x)
* 4 (>10% FO or increase from baseline creatinine of 1.5-1.99x)
* 8 (>15% FO or increase from baseline creatinine of >= 2x).

RAI = Risk score X Injury Score The range of indices is therefore: 1, 2, 3, 4, 5, 6, 8, 10, 12, 20, 24, and 40. RAI >= 8 indicates fulfillment of renal angina ( Basu et al5)

Urine samples: The collection of urine samples is optional for the participating sites. The urine samples will be collected in the morning between 6 and 10 A.M. and/or in the afternoon between 3 and 7 P.M. for up to four days (day 0 through day 3) on all enrolled patients. Some centers may collect daily urine samples, others may choose to collect samples in both time windows. Urine will be drained only from the collection apparatus of an indwelling urinary drainage system or intermittent catheterization. Patients will not be bagged or catheterized separately/independently for the purposes of this study. Collected urine samples will be kept on ice or in 4° C refrigerator until they are processed. During processing, specimens will be centrifuged at 4°C for fifteen minutes. The supernatant will then be divided into up to nine 1-mL aliquots depending on the collected urine volume and stored at minus 80°C. The stored urine samples from all participating sites will be shipped to the Center for Acute Care Nephrology Biomarker Core Laboratory in the Division of Nephrology and Hypertension at Cincinnati Children's Hospital Medical Center when the coordinating site request the samples to be shipped at the time point set forth by the coordinating site. The shipping supplies and instructions will be provided by the coordinating site.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 90 days
* Age less than 25 years

Exclusion Criteria:

* Patients on maintenance hemodialysis, peritoneal dialysis, or with chronic kidney disease with a baseline eGFR of <15 mL/min/1.73m2
* Patients with renal transplant received less than 90 days from the ICU admission.
* Patients admitted to ICU immediately post-operative to within three months following surgical correction of congenital heart disease.
* Patients with uncorrected congenital heart disease. This criteria does not include patients with isolated uncorrected ventricular septal defect (VSD), atrial septal defect (ASD), patent ductus arteriosus (PDA) and patent foramen ovale (PFO).
* Patients following cardiac catheterization.

Ages: 3 Months to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: All medical and surgical patients admitted to the pediatric intensive care unit
Sampling Method: Non-Probability Sample
Enrollment: 5237 (Actual)
Dates: Start 2014-01; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Severe AKI in first seven days of ICU Admission | Within 7 Days of ICU admission
  AKI as defined by KDIGO stage 2 or 3 (by either changes in creatinine or UOP) assessed within 7 days of ICU admission

SECONDARY OUTCOMES:
AKI Conferred Risk on Mortality | 28 days
  After adjustment for covariates, will analyze the independent conferred risk on mortality within 28 days of severe AKI (detected within the first seven days of ICU admission).
Comparison of AKI by Creatinine and Urine Output | 7 and 28 days
  Epidemiology and AKI outcomes for patients will be separated into diagnosis by changes in creatinine, urine output, or both. Independent associations with AKI diagnosed by urine output and outcome will be identified.
Determination of AKI Progression | 7 days
  The stage by stage increase or decrease in AKI severity will be followed - with associations determined - to identify risk factors for AKI progression to severe injury.
Identification of Predictors of Severe AKI | 7 days
  Variables with independent associations for increased risk of severe AKI in the first seven days will be identified.

OTHER OUTCOMES:
Increase in pre-test probability of AKI risk using the renal angina index | 3-4 days
  Assessing all patients with complete data for the presence of renal angina 12 hours after admission using the renal angina index will allow for determination of the heightened prediction of Day 3 - AKI versus standard methods of severity of illness or changes in creatinine alone.
Biomarker incorporation into renal angina index | 3-4 days
  Incorporating values of measured urinary biomarkers, we will determine the additive effect on discriminatory precision for the renal angina index on prediction of Day 3 - AKI

CONTACTS AND LOCATIONS:
Overall Officials: Rajit K Basu, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati; Stuart Goldstein, MD, Principal Investigator — Children's Hospital Medical Center, Cincinnati
Locations (32):
- United States (18):
  - University of Alabama, Birmingham, Alabama
  - Stanford University, Palo Alto, California
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale University, New Haven, Connecticut
  - Nemours/Alfred I. duPont Hospital for Children, Wilmington, Delaware
  - Emory University, Atlanta, Georgia
  - University of Iowa, Des Moines, Iowa
  - University of Michigan, Ann Arbor, Michigan
  - Helen DeVos Children's Hospital, Grand Rapids, Michigan
  - Children's Mercy Hospitals and Clinics, Kansas City, Missouri
  - Washington University in St. Louis, St Louis, Missouri
  - University of New Mexico, Albuquerque, New Mexico
  - Cohen Children's Medical Center of NY, New Hyde Park, New York
  - Stony Brook Long Island Children's Hospital, Stony Brook, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas
  - University of Texas MD Anderson Cancer Center, Houston, Texas
  - Virginia Commonwealth University, Richmond, Virginia
- Australia (2):
  - Children's Hospital at Westmead, Westmead, New South Wales
  - The Sydney Children's Hospitals Network, Sydney
- Canada (3):
  - University of Edmonton, Edmonton
  - Montreal Children's/McGill, Montreal
  - University of British Columbia and Children's and Women's Health Center of British Columbia Branch, Vancouver
- Nanjing Children's Hospital, Nanjing, China
- Indonesia (2):
  - Dept of Child Health Cipto Mangunkusumo/University of Indonesia, Jakarta
  - Dept of Child Health Airlangga University/Dr. Soetomo Hospital, Surabaya
- Ospedale Pediatrico Bambino Gesu, Rome, Italy
- Serbia (2):
  - Mother and Child Health Care, Belgrade
  - University Children's Hospital, Belgrade
- University Children's Medical Institute, National University Hospital, Singapore, Singapore
- Seoul National University Children's Hospital, Seoul, South Korea
- King's College Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes
Individual center data will be distributed per patient/location. Sites will not receive data for patients enrolled at other sites. All data will be centrally housed at Cincinnati Children's Hospital.

REFERENCES:
- [Result] Basu RK, Kaddourah A, Terrell T, Mottes T, Arnold P, Jacobs J, Andringa J, Goldstein SL; Prospective Pediatric AKI Research Group (ppAKI). Assessment of Worldwide Acute Kidney Injury, Renal Angina and Epidemiology in critically ill children (AWARE): study protocol for a prospective observational study. BMC Nephrol. 2015 Feb 26;16:24. doi: 10.1186/s12882-015-0016-6. PMID 25882434
- [Result] Basu RK, Kaddourah A, Terrell T, Mottes T, Arnold P, Jacobs J, Andringa J, Armor M, Hayden L, Goldstein SL. Assessment of Worldwide Acute Kidney Injury, Renal Angina and Epidemiology in Critically Ill Children (AWARE): A Prospective Study to Improve Diagnostic Precision. J Clin Trials. 2015;5(3):222. doi: 10.4172/2167-0870.1000222. Epub 2015 Apr 17. PMID 26719818
- [Derived] Selewski DT, Gist KM, Basu RK, Goldstein SL, Zappitelli M, Soranno DE, Mammen C, Sutherland SM, Askenazi DJ, Ricci Z, Akcan-Arikan A, Gorga SM, Gillespie SE, Woroniecki R; Assessment of the Worldwide Acute Kidney Injury, Renal Angina and Epidemiology (AWARE) Investigators. Impact of the Magnitude and Timing of Fluid Overload on Outcomes in Critically Ill Children: A Report From the Multicenter International Assessment of Worldwide Acute Kidney Injury, Renal Angina, and Epidemiology (AWARE) Study. Crit Care Med. 2023 May 1;51(5):606-618. doi: 10.1097/CCM.0000000000005791. Epub 2023 Feb 17. PMID 36821787
- [Derived] Basu RK, Bjornstad EC, Gist KM, Starr M, Khandhar P, Chanchlani R, Krallman KA, Zappitelli M, Askenazi D, Goldstein SL; SPARC Investigators. Acute kidney injury in critically Ill children and young adults with suspected SARS-CoV2 infection. Pediatr Res. 2022 Jun;91(7):1787-1796. doi: 10.1038/s41390-021-01667-4. Epub 2021 Jul 30. PMID 34331019
- [Derived] Ayalon I, Woo JG, Basu RK, Kaddourah A, Goldstein SL, Kaplan JM; AWARE Investigators. Weight as a Risk Factor for Mortality in Critically Ill Patients. Pediatrics. 2020 Aug;146(2):e20192829. doi: 10.1542/peds.2019-2829. Epub 2020 Jul 3. PMID 32620676
- [Derived] Kaddourah A, Basu RK, Bagshaw SM, Goldstein SL; AWARE Investigators. Epidemiology of Acute Kidney Injury in Critically Ill Children and Young Adults. N Engl J Med. 2017 Jan 5;376(1):11-20. doi: 10.1056/NEJMoa1611391. Epub 2016 Nov 18. PMID 27959707